CLINICAL TRIAL: NCT04394416
Title: Randomized Double-Blind Placebo-Controlled Trial on the Safety and Efficacy of Imatinib for Hospitalized Adults With COVID-19
Brief Title: Trial of Imatinib for Hospitalized Adults With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2038GCCC
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: Arm A: Imatinib
  Arm B: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imatinib (Experimental): Imatinib oral 400 mg daily for 14 days.
  Interventions: Drug: Imatinib
- Placebo (Active Comparator): Placebo oral for 14 days
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Imatinib — Therapeutic
  Arms: Imatinib
Drug: Placebo oral tablet — Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized Double-Blind Placebo-Controlled Trial on the Safety and Efficacy of Imatinib for Hospitalized Adults with COVID-19

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an ongoing global pandemic caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), and at present with no approved or proven antiviral treatment.

Imatinib is a tyrosine kinase inhibitor that has been approved for treatment of many hematologic and solid neoplasm. Imatinib is a weak base that compared to the extracellular compartment is enriched over 1000-fold in the lysosome within several hours as a result of its lysosomotropic property. Imatinib as a weak base accumulates in lysosomes resulting in some antiviral activities by lysosomal alkalization required for virus/cell fusion.

Imatinib demonstrates in vitro activity against SARS-CoV viruses. Imatinib inhibit SARS-CoV and MERS-CoV with micromolar EC50s (range, 9.8 to 17.6 μM) with low toxicity. The mechanism of action studies suggested that ABL-1 tyrosine kinase regulates budding or release of poxviruses and Ebola virus, demonstrating that the c-ABL-1 kinase signaling pathways play an important role in the egress of these viruses. It is also reported that kinase signaling may also be important for replication of two members of the Coronaviridae family, SARS-CoV and MERS-CoV. In vivo studies performed in the mouse model of vaccinia virus infection showed that imatinib was effective in blocking dissemination of the virus.

Imatinib has anti-inflammatory activity including its effectiveness in a "two-hit" murine model of acute lung injury (ALI) caused by combined lipopolysaccharide (LPS) and ventilator-induced lung injury (VILI). Imatinib significantly decreased bronchoalveolar lavage protein, total cells, neutrophils, and TNFα levels in mice exposed to LPS plus VILI, indicating that it attenuates ALI in this clinically relevant model. In another experiment, imatinib attenuated ALI when given 4 hours after LPS, suggesting potential efficacy when given after the onset of injury. Overall, these results strongly suggest the therapeutic potential of imatinib against inflammatory vascular leak and a potential role of imatinib combination therapy for patients with acute respiratory distress syndrome (ARDS) on mechanical ventilation.

The investigators hypothesize that addition of imatinib to the best conventional care (BCC) improves the outcome of hospitalized adult patients with COVID-19. This hypothesis is on the bases of 1) intralysosomal entrapment of imatinib will increase endosomal pH and effectively decrease SARS-CoV-2/cell fusion, 2) kinase inhibitory activity of imatinib will interfere with budding/release or replication of SARS-CoV-2, and 3) because of the critical role of mechanical ventilation in the care of patients with ARDS, imatinib will have a significant clinical impact for patients with severe COVID-19 infection in Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria

Patients may be included in the study only if they meet all of the following criteria:

1. Ability to understand and willingness to sign a written informed consent document. Informed consent must be obtained prior to participation in the study. For patients who are too unwell to provide consent such as patients on invasive ventilator or ECMO, Legally Authorized Representative (LAR) can sign the informed consent.
2. Hospitalized patients ≥ 18 years of age
3. Positive RT-PCR assay for SARS-CoV-2 in the respiratory tract sample (oropharyngeal, nasopharyngeal or BAL) by Center for Disease Control or local laboratory within 7 days of randomization.

Exclusion Criteria

Patients meeting any of the following criteria are not eligible for the study:

1. Patients receiving any other investigational agents in a clinical trial. Off-label use of agents such as hydroxychloroquine is not an exclusion criterion. Therapies that are shown to be effective but may not be licensed can be added as an exception to the exclusion criteria in order to allow for the most contemporary standard of care to include emergency use authorization treatments as they become available. Antivirals such as remdesivir will be permissible given the FDA authorized emergency use.
2. Pregnant or breastfeeding women.
3. Patients with significant liver or renal dysfunction function at screen as defined as:

   * Direct bilirubin > 2.5 mg/dL
   * AST, ALT, or alkaline phosphatase > 5 x upper limit of normal
   * eGFR ≤ 30 mL/min or requiring renal replacement therapy
4. Patients with significant hematologic disorder at screen as defined as:

   * Absolute neutrophil count (ANC) < 500/μL
   * Platelet < 20,000/μL
   * Hemoglobin < 7 g/dL
5. Uncontrolled undercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled active seizure disorder, or psychiatric illness/social situations that per site Principal Investigator's judgment would limit compliance with study requirements.
6. Known allergy to imatinib or its component products.
7. Any other clinical conditions that in the opinion of the investigator would make the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a two-point change using the 8-category ordinal scale | Day 14 from baseline
  The ordinal scale is an evaluation of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring supplemental oxygen; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death.

SECONDARY OUTCOMES:
All-Cause mortality | Day 28 and Day 60 post baseline
  All-cause mortality post baseline
Time to a 2-point clinical change | Up to 60 days post baseline
  Time to a 2-point clinical change difference
Hospitalization | Up to 60 days post baseline
  Duration of hospitalization
Duration of ECMO or invasive mechanical ventilation | Up to 60 days post baseline
  For subjects who are on ECMO or mechanical ventilation at Day 1
Duration of ICU stay | Up to 60 days post baseline
  For subjects who are in ICU at Day 1
SARS-CoV-2 negative | Up to 60 days post baseline
  Time to SARS-CoV-2 negative by reverse transcriptase-polymerase chain reaction (RT-PCR)
Negative oropharyngeal or nasopharyngeal swab | Up to 28 days post baseline
  Proportion of patients with negative oropharyngeal or nasopharyngeal swab for SARS-CoV-2 by quantitative RT PCR on days 5, 10, 14, 21, and 28 after starting treatment
Serious adverse events (SAEs) | Up to 60 days post baseline
  Proportion of subjects with serious adverse events
Discontinuation due to adverse events | Up to 60 days post baseline
  Proportion of subjects who discontinue study drug due to adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Liu K, Fang YY, Deng Y, Liu W, Wang MF, Ma JP, Xiao W, Wang YN, Zhong MH, Li CH, Li GC, Liu HG. Clinical characteristics of novel coronavirus cases in tertiary hospitals in Hubei Province. Chin Med J (Engl). 2020 May 5;133(9):1025-1031. doi: 10.1097/CM9.0000000000000744. PMID 32044814
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Al-Bari MA. Chloroquine analogues in drug discovery: new directions of uses, mechanisms of actions and toxic manifestations from malaria to multifarious diseases. J Antimicrob Chemother. 2015;70(6):1608-21. doi: 10.1093/jac/dkv018. Epub 2015 Feb 17. PMID 25693996
- [Background] Daniel WA, Bickel MH, Honegger UE. The contribution of lysosomal trapping in the uptake of desipramine and chloroquine by different tissues. Pharmacol Toxicol. 1995 Dec;77(6):402-6. doi: 10.1111/j.1600-0773.1995.tb01050.x. PMID 8835367
- [Background] Savarino A, Boelaert JR, Cassone A, Majori G, Cauda R. Effects of chloroquine on viral infections: an old drug against today's diseases? Lancet Infect Dis. 2003 Nov;3(11):722-7. doi: 10.1016/s1473-3099(03)00806-5. PMID 14592603
- [Background] Yan Y, Zou Z, Sun Y, Li X, Xu KF, Wei Y, Jin N, Jiang C. Anti-malaria drug chloroquine is highly effective in treating avian influenza A H5N1 virus infection in an animal model. Cell Res. 2013 Feb;23(2):300-2. doi: 10.1038/cr.2012.165. Epub 2012 Dec 4. No abstract available. PMID 23208422
- [Background] Keyaerts E, Vijgen L, Maes P, Neyts J, Van Ranst M. In vitro inhibition of severe acute respiratory syndrome coronavirus by chloroquine. Biochem Biophys Res Commun. 2004 Oct 8;323(1):264-8. doi: 10.1016/j.bbrc.2004.08.085. PMID 15351731
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Biot C, Daher W, Chavain N, Fandeur T, Khalife J, Dive D, De Clercq E. Design and synthesis of hydroxyferroquine derivatives with antimalarial and antiviral activities. J Med Chem. 2006 May 4;49(9):2845-9. doi: 10.1021/jm0601856. PMID 16640347
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Chapuy B, Panse M, Radunski U, Koch R, Wenzel D, Inagaki N, Haase D, Truemper L, Wulf GG. ABC transporter A3 facilitates lysosomal sequestration of imatinib and modulates susceptibility of chronic myeloid leukemia cell lines to this drug. Haematologica. 2009 Nov;94(11):1528-36. doi: 10.3324/haematol.2009.008631. PMID 19880777
- [Background] Gotink KJ, Broxterman HJ, Labots M, de Haas RR, Dekker H, Honeywell RJ, Rudek MA, Beerepoot LV, Musters RJ, Jansen G, Griffioen AW, Assaraf YG, Pili R, Peters GJ, Verheul HM. Lysosomal sequestration of sunitinib: a novel mechanism of drug resistance. Clin Cancer Res. 2011 Dec 1;17(23):7337-46. doi: 10.1158/1078-0432.CCR-11-1667. Epub 2011 Oct 6. PMID 21980135
- [Background] Gotink KJ, Rovithi M, de Haas RR, Honeywell RJ, Dekker H, Poel D, Azijli K, Peters GJ, Broxterman HJ, Verheul HM. Cross-resistance to clinically used tyrosine kinase inhibitors sunitinib, sorafenib and pazopanib. Cell Oncol (Dordr). 2015 Apr;38(2):119-29. doi: 10.1007/s13402-015-0218-8. Epub 2015 Feb 11. PMID 25665527
- [Background] Colombo F, Trombetta E, Cetrangolo P, Maggioni M, Razini P, De Santis F, Torrente Y, Prati D, Torresani E, Porretti L. Giant Lysosomes as a Chemotherapy Resistance Mechanism in Hepatocellular Carcinoma Cells. PLoS One. 2014 Dec 10;9(12):e114787. doi: 10.1371/journal.pone.0114787. eCollection 2014. PMID 25493932
- [Background] Ruzickova E, Skoupa N, Dolezel P, Smith DA, Mlejnek P. The Lysosomal Sequestration of Tyrosine Kinase Inhibitors and Drug Resistance. Biomolecules. 2019 Oct 31;9(11):675. doi: 10.3390/biom9110675. PMID 31683643
- [Background] Burger H, den Dekker AT, Segeletz S, Boersma AW, de Bruijn P, Debiec-Rychter M, Taguchi T, Sleijfer S, Sparreboom A, Mathijssen RH, Wiemer EA. Lysosomal Sequestration Determines Intracellular Imatinib Levels. Mol Pharmacol. 2015 Sep;88(3):477-87. doi: 10.1124/mol.114.097451. Epub 2015 Jun 24. PMID 26108972
- [Background] Fu D, Zhou J, Zhu WS, Manley PW, Wang YK, Hood T, Wylie A, Xie XS. Imaging the intracellular distribution of tyrosine kinase inhibitors in living cells with quantitative hyperspectral stimulated Raman scattering. Nat Chem. 2014 Jul;6(7):614-22. doi: 10.1038/nchem.1961. Epub 2014 May 25. PMID 24950332
- [Background] Chilakapati SR, Serasanambati M, Vissavajjhala P, Kanala JR, Chilakapati DR. Amelioration of bleomycin-induced pulmonary fibrosis in a mouse model by a combination therapy of bosentan and imatinib. Exp Lung Res. 2015 May;41(4):173-88. doi: 10.3109/01902148.2014.939312. Epub 2015 Apr 6. PMID 25844688
- [Background] Li M, Abdollahi A, Grone HJ, Lipson KE, Belka C, Huber PE. Late treatment with imatinib mesylate ameliorates radiation-induced lung fibrosis in a mouse model. Radiat Oncol. 2009 Dec 21;4:66. doi: 10.1186/1748-717X-4-66. PMID 20025728
- [Background] Wolf AM, Wolf D, Rumpold H, Ludwiczek S, Enrich B, Gastl G, Weiss G, Tilg H. The kinase inhibitor imatinib mesylate inhibits TNF-alpha production in vitro and prevents TNF-dependent acute hepatic inflammation. Proc Natl Acad Sci U S A. 2005 Sep 20;102(38):13622-7. doi: 10.1073/pnas.0501758102. Epub 2005 Sep 8. PMID 16174751
- [Background] Rizzo AN, Sammani S, Esquinca AE, Jacobson JR, Garcia JG, Letsiou E, Dudek SM. Imatinib attenuates inflammation and vascular leak in a clinically relevant two-hit model of acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2015 Dec 1;309(11):L1294-304. doi: 10.1152/ajplung.00031.2015. Epub 2015 Oct 2. PMID 26432864
- [Background] Schrezenmeier E, Dorner T. Mechanisms of action of hydroxychloroquine and chloroquine: implications for rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):155-166. doi: 10.1038/s41584-020-0372-x. Epub 2020 Feb 7. PMID 32034323
- [Background] Horne GA, Stobo J, Kelly C, Mukhopadhyay A, Latif AL, Dixon-Hughes J, McMahon L, Cony-Makhoul P, Byrne J, Smith G, Koschmieder S, BrUmmendorf TH, Schafhausen P, Gallipoli P, Thomson F, Cong W, Clark RE, Milojkovic D, Helgason GV, Foroni L, Nicolini FE, Holyoake TL, Copland M. A randomised phase II trial of hydroxychloroquine and imatinib versus imatinib alone for patients with chronic myeloid leukaemia in major cytogenetic response with residual disease. Leukemia. 2020 Jul;34(7):1775-1786. doi: 10.1038/s41375-019-0700-9. Epub 2020 Jan 10. PMID 31925317
- [Background] Wang Y, Fan G, Salam A, Horby P, Hayden FG, Chen C, Pan J, Zheng J, Lu B, Guo L, Wang C, Cao B. Comparative Effectiveness of Combined Favipiravir and Oseltamivir Therapy Versus Oseltamivir Monotherapy in Critically Ill Patients With Influenza Virus Infection. J Infect Dis. 2020 Apr 27;221(10):1688-1698. doi: 10.1093/infdis/jiz656. PMID 31822885
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Rainsford KD, Parke AL, Clifford-Rashotte M, Kean WF. Therapy and pharmacological properties of hydroxychloroquine and chloroquine in treatment of systemic lupus erythematosus, rheumatoid arthritis and related diseases. Inflammopharmacology. 2015 Oct;23(5):231-69. doi: 10.1007/s10787-015-0239-y. Epub 2015 Aug 6. PMID 26246395
- [Background] Cutler DJ, MacIntyre AC, Tett SE. Pharmacokinetics and cellular uptake of 4-aminoquinoline antimalarials. Agents Actions Suppl. 1988;24:142-57. doi: 10.1007/978-3-0348-9160-8_13. No abstract available. PMID 3263755
- [Background] Tett SE. Clinical pharmacokinetics of slow-acting antirheumatic drugs. Clin Pharmacokinet. 1993 Nov;25(5):392-407. doi: 10.2165/00003088-199325050-00005. PMID 7904547
- [Background] Carmichael SJ, Charles B, Tett SE. Population pharmacokinetics of hydroxychloroquine in patients with rheumatoid arthritis. Ther Drug Monit. 2003 Dec;25(6):671-81. doi: 10.1097/00007691-200312000-00005. PMID 14639053
- [Background] Yusuf IH, Foot B, Galloway J, Ardern-Jones MR, Watson SL, Yelf C, Burdon MA, Bishop PN, Lotery AJ. The Royal College of Ophthalmologists recommendations on screening for hydroxychloroquine and chloroquine users in the United Kingdom: executive summary. Eye (Lond). 2018 Jul;32(7):1168-1173. doi: 10.1038/s41433-018-0136-x. Epub 2018 Jun 11. No abstract available. PMID 29887605
- [Background] Chatre C, Roubille F, Vernhet H, Jorgensen C, Pers YM. Cardiac Complications Attributed to Chloroquine and Hydroxychloroquine: A Systematic Review of the Literature. Drug Saf. 2018 Oct;41(10):919-931. doi: 10.1007/s40264-018-0689-4. PMID 29858838
- [Background] McHenry AR, Wempe MF, Rice PJ. Stability of Extemporaneously Prepared Hydroxychloroquine Sulfate 25-mg/mL Suspensions in Plastic Bottles and Syringes. Int J Pharm Compd. 2017 May-Jun;21(3):251-254. PMID 28557788
- [Derived] Emadi A, Chua JV, Talwani R, Bentzen SM, Baddley J. Safety and Efficacy of Imatinib for Hospitalized Adults with COVID-19: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 28;21(1):897. doi: 10.1186/s13063-020-04819-9. PMID 33115543
- [Derived] Zhao H, Mendenhall M, Deininger MW. Imatinib is not a potent anti-SARS-CoV-2 drug. Leukemia. 2020 Nov;34(11):3085-3087. doi: 10.1038/s41375-020-01045-9. Epub 2020 Sep 30. No abstract available. PMID 32999432
- See also: FDA. Imatinib Label. Food and Drug Administration 2018 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/021588s053lbl.pdf
- See also: WHO. Coronavirus disease (COVID-2019) R&D Blueprint. World Health Organization 2020 — http://www.who.int/blueprint/priority-diseases/key-action/novel-coronavirus/en/